CLINICAL TRIAL: NCT03005730
Title: Influence of Photobiomodulation In The Masseter and Temporal On Pain, Joint Mobility In Individuals With Temporomandibular Joint Dysfunction: Clinical Trial Randomised, Placebo-Controlled And Double-Blind
Brief Title: Photobiomodulation In the Masseter and Temporal In Patients With Temporomandibular Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Daniela Ap. Biasotto-Gonzalez, Doctor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHOTOBIOMODULATION DTM EXT.
Record Dates: First submitted 2016-12-26; First posted 2016-12-29 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Temporomandibular Disorder
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Experimental): Submitted to a session of phototherapy with 39,27 Joules per point in muscle masseter and temporal bilateral.
  Interventions: Other: phototherapy
- Group 2 (Placebo Comparator): Submitted to a session of phototherapy placebo with 0,0 Joules per point in muscle masseter and temporal bilateral.
  Interventions: Other: phototherapy placebo

INTERVENTIONS:
Other: phototherapy — The portable PainAway® nine-diode cluster (Multi Radiance Medical®, Solon, OH, USA) will be employed. This system has one 905 nm laser diode, four 875 nm LED diodes and four 670 nm LED diodes. The aperture size of device is 4 cm2.
  Arms: Group 1
Other: phototherapy placebo — The placebo portable. The aperture size of device is 4 cm2 .
  Arms: Group 2

SUMMARY:
Background: According to the International Association for the Study of Pain (IASP), the term temporomandibular disorder (TMD) regards a subgroup of orofacial pain, the symptoms of which include pain or discomfort in the temporomandibular joint, ears, masticatory muscles and neck on one or both sides as well as joint sounds, limited mandibular movements or mandibular deviation and difficulties chewing. Phototherapy, such as low level laser therapy (LLLT) and light-emitting diode (LED) therapy, is one of the resources used to treatment muscle pain. Thus, there is a need to investigate therapeutic resources that combine different wavelengths as well as different light sources (LLLT and LED) in the same apparatus.

Question: The aim of the proposed study is to evaluate the effects of phototherapy on pain, activity of the masticatory muscles (masseter and anterior temporal bilaterally) and joint mobility in individuals with temporomandibular disorder (TMD). A further aim is to determine the cumulative effect 24 and 48 hours after a six session.

Methods/Design: A placebo-controlled, double-blind, randomized, clinical trial will be carried out involving 30 women between 18 and 40 years of age with a diagnosis of myogenous TMD. The participants will then be randomly allocated to two groups totaling 15 individuals per group. Group 1 submitted to a session of phototherapy with 39,27 Joules per point one group will receive placebo therapy (0 Joules). The following assessment tools will be administered on four separate occasions (baseline and immediately after, 24 h after and 48 h after phototherapy). Pain intensity will be assessed using the visual analog scale for pain, meter for range of movement, and electromyographic EMG analysis on the masseter and anterior temporal muscles.

Discussion: The study will support the practice of evidence-based to the use of phototherapy in individuals with a myogenous TMD. Data will be published after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

* All volunteers will have a diagnosis of myogenous TMD based on the RDC/TMD with moderate to severe pain in the masseter and temporal muscles rated by an expert dentist. To standardize the sample, the body mass index of all participants must be less than 25 kg/m2, as the amount of adipose tissue between the electrode and surface of the muscle can affect that reading of the electromyographic (EMG) signal. All volunteers must also have an initial pain score greater than 3 points on the VAS.

Exclusion Criteria:

* The exclusion criteria will be missing teeth, the use of dentures, systemic or neuromuscular diseases, a history of trauma to the face or temporomandibular joint, history of temporomandibular joint luxation, currently undergoing orthodontic treatment, or currently undergoing medicinal treatment that can affect the musculoskeletal system (analgesic, anti-inflammatory agent or muscle relaxant).

Ages: 1 Year to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2016-12-10 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2018-01-20 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 5 min
  A Visual analog scale allows the quantification of pain intensity. This scale consists of a straight line measuring 10 cm in length, with "absence of pain" written at one end and "worst pain ever felt" written at the other end. The volunteer will be instructed to make a perpendicular line between the two extremes that represents the pain level he/she is feeling at the time

SECONDARY OUTCOMES:
Range of motion | 10 min
  We used a Starrett digital caliper ® to assess the breadth of mandibular movement (in mm), that is, the opening of the mouth was measured according to the RDC/TMD, and right and left lateral excursions.